CLINICAL TRIAL: NCT06821555
Title: Pengembangan Model Mindful Eating Intervention Dengan Aplikasi (EATS UP) Pada Remaja Obes Dan Pengaruhnya Terhadap Komposisi Tubuh Dan Resistensi Insulin (Indonesia Language)
Brief Title: Mindful Eating Intervention Using EATS UP App: Effects on Body Composition and Insulin Resistance in Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aryono Hendarto, Professor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-07-1125
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Adolescent Obesity; Eating Behaviors; Nutrition Status; Blood Glucose; Body Fat Composition
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutrition and Physical Activity with Mindful Eating Intervention (Experimental): The intervention group receiving nutrition and physical activity with mindful eating intervention
  Interventions: Behavioral: Nutrition and Physical Activity Education with Mindful Eating Intervention
- Nutrition and Physical Activity Education (Experimental): The control group receiving only nutrition and physical activity education
  Interventions: Behavioral: Nutrition and Physical Activity Education

INTERVENTIONS:
Behavioral: Nutrition and Physical Activity Education with Mindful Eating Intervention — Mindful Eating Intervention applied to Obesity treatment for Adolescent alongside with Nutrition and Physical Activity Education from Nutritionist and Psychologist
  Arms: Nutrition and Physical Activity with Mindful Eating Intervention
Behavioral: Nutrition and Physical Activity Education — Nutrition and physical activity education from Nutritionist applied as Obesity treatment for Adolescent
  Arms: Nutrition and Physical Activity Education

SUMMARY:
The goal of this experimental study is to develop and evaluate the effectiveness of a Mindful Eating Intervention (MEI) model integrated with the digital application EatsUp for improving body fat percentage among obese adolescents in Indonesia. The study aims to address the rising prevalence of adolescent obesity and its associated health risks, such as insulin resistance and cardiometabolic syndrome, by promoting mindful eating habits and healthy lifestyle behaviors.

The main questions it aims to answer are:

* Is the MEI model valid and acceptable for use among obese adolescents?
* Does the MEI model reduce:

  * Body fat percentage?
  * Waist-to-height ratio (WHtR)?
  * Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)?
* Does the MEI model improve eating behavior scores compared to a control group over 12 weeks?

Participants will:

* Use the EatsUp app, designed to monitor calorie intake/output and deliver mindful eating and nutrition education.
* Receive training on mindfulness-based eating practices, along with guidance on balanced nutrition and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15-18 years old
* Agreed to be involved in research proven by signing informed consent and assent
* Indicated as Obesity by BMI-Age Nutritional Status and body fat percentage

Exclusion Criteria:

* Subject is on a dietary treatment or has a serious condition (e.g. chronic infectious disease, and undergoing drug therapy)
* Subject with special needs (cannot use internet, cannot communicate normally)

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Body Composition | From enrollment to the end of intervention at 12 weeks
  Body composition measured in this study are Body Mass Index for Age (BMI-Age), Waist-to-Height Ratio (WHtR), Waist Circumference, Body Fat Percentage,
Fasting Blood Sugar Levels | From enrollment to the end of intervention at 12 weeks
  Blood glucose examination is carried out after fasting for 10 - 12 hours.
Fasting Insulin Levels | From enrollment to the end of intervention at 12 weeks
  Measures the amount of insulin in the blood during fasting.
Insulin Resistance | From enrollment to the end of intervention at 12 weeks
  HOMA-IR (Homeostatic Model Assessment for Insulin Resistance): Calculated using fasting glucose and insulin levels, with a threshold value (≥3.8) indicating insulin resistance.
Mindful Eating Score | From enrollment to the end of intervention at 12 weeks
  Mindful eating is assessed based on 5 domains: distraction, disinhibition, awareness, external cues, and emotional eating. Mindful Eating Questionnaire is scored by adding up responses to each item and dividing by the total number of items answered. The resulting score ranges from 1 to 4, with higher scores indicating more mindful eating.
Eating Behavior | From enrollment to the end of intervention at 12 weeks
  Psychosocial factors and attitudes that influence eating behavior such as food choices, dieting, and the presence of eating disorders measured using Adolescent Food Habit Checklist (AFHC)
Binge Eating | From enrollment to the end of intervention at 12 weeks
  Eating behavior disorder where a person tends to overeat and has difficulty controlling it is assessed from a total score of 16 statements using Binge Eating Scale Questionnaire. The total score ranges from 0 to 46, with higher scores correlating with more frequent and severe binge eating behaviors. Based on the total scores, it can be classified into distinct severity categories as follows:
  1. Low Binge-Eating: Scores of 17 or lower;
  2. Mild to Moderate Binge-Eating: Scores ranging from 18 to 26;
  3. Severe Binge-Eating: Scores of 27 or higher, indicating a high frequency and severity of binge-eating symptoms.
Sleep Quality | From enrollment to the end of intervention at 12 weeks
  Sleep can produce a feeling of being fit, assessed based on duration, latency, efficiency and sleep disturbance as measured using the Pittsburgh Sleep Quality Index (PSQI) questionnaire.
Physical Activity Level | From enrollment to the end of intervention at 12 weeks
  Measurement of physical activity during the last 7 days using the International Physical Activity Questionnaire for Adolescent (IPAQ-A)

CONTACTS AND LOCATIONS:
Overall Officials: Aryono Hendarto, PhD, Principal Investigator — Indonesia University
Locations (1):
- Universitas Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No